CLINICAL TRIAL: NCT05310409
Title: A Prospective Cohort Study Evaluating PAN-PROMISE, a Patient-Reported Outcome Measure, To Detect and Risk-Stratify Post-ERCP Pancreatitis
Brief Title: PAN-PROMISE to Detect Post-ERCP Pancreatitis Symptoms
Acronym: PAN-PROMISE
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: PAN-PROMISE
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Post-ERCP Acute Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to use a validated patient-reported outcome measure to evaluate how many patients have symptoms of pancreatitis after ERCP and how it correlates with their quality of life and productivity.

DETAILED DESCRIPTION:
This project will measure the impact of a recently validated patient-reported outcome measure for acute pancreatitis, PAN-PROMISE, to detect post-ERCP pancreatitis symptoms and capture its morbidity. The study will compare the change of PAN-PROMISE before and after ERCP to the current standard diagnostic criteria for post-ERCP pancreatitis, the Cotton Consensus Criteria. The main limitations of the Cotton-Consensus Criteria are that it fails to capture outpatient or ambulatory morbidity, uses length of stay to define the severity of pancreatitis without accounting for local or systemic complications for pancreatitis, and it has limited sensitivity in patients with chronic symptoms such as patients with chronic pancreatitis or pancreatic adenocarcinoma. These limitations have impeded the evaluation of potential therapies to prevent post-ERCP pancreatitis. PAN-PROMISE will help capture and quantitate the morbidity related to post-ERCP pancreatitis and thus will enhance our ability to optimize outcomes following ERCP.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing ERCP
2. Age >= 18 years old
3. Intact major papilla

Exclusion Criteria:

1. Unwillingness or inability to consent for the study
2. Age < 18 years
3. Standard contraindications to ERCP
4. Intrauterine pregnancy
5. Prior hepaticojejunostomy in a patient undergoing ERCP for a bile duct indication
6. Prior pancreaticojejunostomy in a patient undergoing ERCP for a pancreatic duct indication
7. Low probability of completing the follow-up
8. Acute pancreatitis (by the Revised Atlanta criteria) in the seven days prior to ERCP.
9. Patients who do not answer at least 80% of the questions on the baseline and 48-hour follow-up survey.
10. Patients who could not be contacted via a telephone call to assess for post-ERCP complications at 48-72 hours.
11. Patients who speak a language other than English, Spanish, Bulgarian, Mandarin, English, French, German, Greek, Hungarian, Italian, Korean, Polish, Portuguese, Romanian, Russian, Turkish, Ukrainian, or Hindi (as the PAN-PROMISE has only been translated and validated in these languages.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We are enrolling patients who are undergoing ERCP at our two centers.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Post-ERCP Pancreatitis | 7 days after ERCP
  will define post-ERCP pancreatitis using the Cotton Consensus Criteria with a 3 physician adjudication committee.
PROM-PEP | 30 days
  will capture the work abseentism and loss of productivity using the Work-Productivity and Activity Impairment Questionnaire and will express in in 2021 US Dollars.

SECONDARY OUTCOMES:
Direct Health Care Costs | 30 days
  will capture the direct healthcare costs using the Medicare Reimbursement data and express it in 2021 US Dollars.

OTHER OUTCOMES:
Quality of Life Assessment | 30 days
  will capture changes in Quality of Life using the SF-12 instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Kochman, MD, Principal Investigator — University of Pennsylvania; Mustafa Arain, MD, Principal Investigator — University of California, San Francisco; Nikhil R Thiruvengadam, MD, Principal Investigator — Loma Linda University School of Medicine.
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Masci E, Toti G, Mariani A, Curioni S, Lomazzi A, Dinelli M, Minoli G, Crosta C, Comin U, Fertitta A, Prada A, Passoni GR, Testoni PA. Complications of diagnostic and therapeutic ERCP: a prospective multicenter study. Am J Gastroenterol. 2001 Feb;96(2):417-23. doi: 10.1111/j.1572-0241.2001.03594.x. PMID 11232684
- [Background] Artifon EL, Chu A, Freeman M, Sakai P, Usmani A, Kumar A. A comparison of the consensus and clinical definitions of pancreatitis with a proposal to redefine post-endoscopic retrograde cholangiopancreatography pancreatitis. Pancreas. 2010 May;39(4):530-5. doi: 10.1097/MPA.0b013e3181c306c0. PMID 20093992
- [Background] Thiruvengadam NR, Forde KA, Ma GK, Ahmad N, Chandrasekhara V, Ginsberg GG, Ho IK, Jaffe D, Panganamamula KV, Kochman ML. Rectal Indomethacin Reduces Pancreatitis in High- and Low-Risk Patients Undergoing Endoscopic Retrograde Cholangiopancreatography. Gastroenterology. 2016 Aug;151(2):288-297.e4. doi: 10.1053/j.gastro.2016.04.048. Epub 2016 May 20. PMID 27215656
- [Background] de-Madaria E, Sanchez-Marin C, Carrillo I, Vege SS, Chooklin S, Bilyak A, Mejuto R, Mauriz V, Hegyi P, Marta K, Kamal A, Lauret-Brana E, Barbu ST, Nunes V, Ruiz-Rebollo ML, Garcia-Rayado G, Lozada-Hernandez EE, Pereira J, Negoi I, Espina S, Hollenbach M, Litvin A, Bolado-Concejo F, Vargas RD, Pascual-Moreno I, Singh VK, Mira JJ. Design and validation of a patient-reported outcome measure scale in acute pancreatitis: the PAN-PROMISE study. Gut. 2021 Jan;70(1):139-147. doi: 10.1136/gutjnl-2020-320729. Epub 2020 Apr 3. PMID 32245906
- [Derived] Thiruvengadam NR, Kouanda A, Kalluri A, Schaubel D, Saumoy M, Forde K, Song J, Faggen A, Davis BG, Onwugaje KC, Cote G, Arain MA, Kochman ML. A Prospective Cohort Study Evaluating PAN-PROMISE, a Patient-reported Outcome Measure to Detect Post-ERCP Morbidity. Clin Gastroenterol Hepatol. 2023 May;21(5):1233-1242.e14. doi: 10.1016/j.cgh.2022.08.034. Epub 2022 Sep 6. PMID 36075501